CLINICAL TRIAL: NCT01680640
Title: Investigation of the Effects of a Synbiotic on Liver Fat, Disease Biomarkers and Intestinal Microbiota in Non-alcoholic Fatty Liver Disease
Brief Title: Investigation of Synbiotic Treatment in NAFLD
Acronym: INSYTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RHM MED1071
Record Dates: First submitted 2012-08-24; First posted 2012-09-07 (Estimated); Results first posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2020-10

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: non alcoholic fatty liver disease; NAFLD; synbiotic; gut microbiota; intervention; RCT (Randomized Clinical Trial); biomarkers
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Synbiotics; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Synbiotic (Active Comparator): Fructo-oligosacharide with a degree of polymerization < 10 at 4 g/twice a day (two sticks a day) plus Bifidobacterium animalis subsp. lactis (BB-12) as minimum of 10 billion colony forming unit (CFU)/day (1 capsule a day).
  Interventions: Dietary Supplement: Synbiotic
- Maltodextrin (Placebo Comparator): 4 grams of maltodextrin daily.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Synbiotic — The synbiotic to be used is fructo-oligosacharide with a degree of polymerization < 10 at 4 g/twice a day (two sticks a day) plus Bifidobacterium animalis subsp. lactis BB-12 as minimum of 10 billion CFU/day (1 capsule a day).
  Arms: Synbiotic
Dietary Supplement: Maltodextrin
  Arms: Maltodextrin

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is a liver condition in which fat builds up in the liver not caused by alcohol. The liver is an organ that is not designed to build up fat. NAFLD is common in people who have too much body fat in their abdomen or who have diabetes (high blood sugar), but does not always exist with these conditions. NAFLD can also occur in thin people too. NAFLD can be harmful to the liver and may cause the liver to fail over time. NAFLD may also cause adult (or type 2) diabetes and also heart disease. In people who already have diabetes, NAFLD can cause glucose (sugar) levels to be too high.

Our intestines (guts) contain healthy bacteria and some harmful bacteria (bugs). This balance of healthy and harmful bugs is essential for the normal workings of our intestine to digest food. Providing these bacteria do not leak out into the blood they do not cause harm. If the balance of healthy to harmful bugs is upset, the harmful can cause problems and leak out into the blood. Because the liver is connected to the intestine by blood vessels the harmful bacteria can get to the liver and cause problems. These bacteria can cause the liver and the body to build up too much fat and might cause NAFLD and obesity. In this study, we will test the effects of a supplement (synbiotic) taken during the day, that contains a mixture of 'good' healthy bacteria (probiotic) and a sugar (prebiotic) that is not broken down and absorbed into the blood. We will test whether the synbiotic supplement has beneficial effects on the NAFLD liver condition and on factors linked to too much body fat, diabetes and heart disease.

DETAILED DESCRIPTION:
We will recruit people with NAFLD who have been diagnosed as part of their NHS (National Health Service) care with having this condition. At present there is no treatment for this condition.

Purpose and design:

We are asking the research question: "Does the modulation of gut microflora with a synbiotic improve non-alcoholic fatty liver disease and the related risk factors for heart disease and type 2 diabetes?"

Presently there is no treatment for this liver condition. Research evidence suggests that a synbiotic supplement might be beneficial for this condition.

To address this research question we want to undertake a randomised double blind placebo controlled trial recruiting people who have been diagnosed with NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* Both men and women
* Age > 18 years
* Liver fat diagnosed on normal clinical grounds including in most cases liver assessed by Kleiner scoring system to classify severity, with no known aetiological factors for underlying liver disease (e.g. exclusion of hepatitis A, B & C, primary biliary cirrhosis, autoimmune hepatitis, haemochromatosis). Last liver biopsy will be within 3 years of recruitment to the study.
* Liver fat diagnosed by ultrasound, CT or magnetic resonance imaging (MRI) in patients who also have either diabetes and/or features of the metabolic syndrome, without evidence of known aetiological factors for underlying liver disease (e.g. exclusion of hepatitis A, B & C, primary biliary cirrhosis, autoimmune hepatitis, haemochromatosis).
* Alcohol consumption ≤ 14 units / week for women ≤ 21 units / week for men.

Exclusion Criteria:

* Alcohol consumption > 15 units /week for women and > 22 units /week for men.
* Decompensated acute or chronic liver disease.
* A history of viral hepatitis, diarrhoea, diverticulosis, irritable bowel syndrome, inflammatory bowel diseases, coeliac disease (seropositivity for anti-endomysial immunoglobulin A antibodies; immunoglobulin A (IgA) EMA).
* Previous bariatric or other abdominal surgery.
* Continuous use of antibiotics that may change gut microflora, probiotics, or antisecretory drugs capable of causing achlorhydria within the 2 months preceding enrolment, or evidence of immunoglobulin A or immunoglobulin deficiency (both of which produce confounding effects during assessments of intestinal permeability and small intestinal bacterial overgrowth).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2013-12; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Byrne, MBBCh, PhD, Principal Investigator — University of Southampton/University Hospital Southampton NHS Foundation Trust
Locations (1):
- Southamption General Hospital, Southampton, Hants, United Kingdom

REFERENCES:
- [Derived] Scorletti E, Afolabi PR, Miles EA, Smith DE, Almehmadi A, Alshathry A, Childs CE, Del Fabbro S, Bilson J, Moyses HE, Clough GF, Sethi JK, Patel J, Wright M, Breen DJ, Peebles C, Darekar A, Aspinall R, Fowell AJ, Dowman JK, Nobili V, Targher G, Delzenne NM, Bindels LB, Calder PC, Byrne CD. Synbiotics Alter Fecal Microbiomes, But Not Liver Fat or Fibrosis, in a Randomized Trial of Patients With Nonalcoholic Fatty Liver Disease. Gastroenterology. 2020 May;158(6):1597-1610.e7. doi: 10.1053/j.gastro.2020.01.031. Epub 2020 Jan 25. PMID 31987796
- [Derived] Scorletti E, Afolabi PR, Miles EA, Smith DE, Almehmadi A, Alshathry A, Moyses HE, Clough GF, Wright M, Patel J, Bindels L, Delzenne NM, Calder PC, Byrne CD. Design and rationale of the INSYTE study: A randomised, placebo controlled study to test the efficacy of a synbiotic on liver fat, disease biomarkers and intestinal microbiota in non-alcoholic fatty liver disease. Contemp Clin Trials. 2018 Aug;71:113-123. doi: 10.1016/j.cct.2018.05.010. Epub 2018 May 19. PMID 29787859
- [Derived] Byrne CD, Targher G. Time to Replace Assessment of Liver Histology With MR-Based Imaging Tests to Assess Efficacy of Interventions for Nonalcoholic Fatty Liver Disease. Gastroenterology. 2016 Jan;150(1):7-10. doi: 10.1053/j.gastro.2015.11.016. Epub 2015 Nov 18. No abstract available. PMID 26602219
- [Derived] Byrne CD, Targher G. Ectopic fat, insulin resistance, and nonalcoholic fatty liver disease: implications for cardiovascular disease. Arterioscler Thromb Vasc Biol. 2014 Jun;34(6):1155-61. doi: 10.1161/ATVBAHA.114.303034. Epub 2014 Apr 17. PMID 24743428

RESULTS

PARTICIPANT FLOW:
Groups:
- Synbiotic: Fructo-oligosaccharide with a degree of polymerization < 10 at 4 g/twice a day (two sticks a day) plus Bifidobacterium animalis subsp. lactis BB-12 as minimum of 10 billion CFU/day (1 capsule a day).
  Synbiotic: The synbiotic to be used is fructo-oligosachharide with a degree of polymerization < 10 at 4 g/twice a day (two sticks a day) plus Bifidobacterium animalis subsp. lactis BB-12 as minimum of 10 billion CFU/day (1 capsule a day).
- Maltodextrin: 4 grams of maltodextrin daily.
  Maltodextrin
Period: Overall Study
Arm/Group | Synbiotic | Maltodextrin
Started | 55 | 49
Completed | 45 | 44
Not Completed | 10 | 5

BASELINE CHARACTERISTICS:
Population: The ITT analysis included all patients randomized who had baseline and end-of-study measurements, regardless of whether they were later found to be ineligible, a protocol violator, given the wrong treatment allocation, or never treated.
Groups:
- Synbiotic: Fructo-oligosaccharide with a degree of polymerization < 10 at 4 g/twice a day (two sticks a day) plus Bifidobacterium animalis subsp. lactis BB-12 as minimum of 10 billion CFU/day (1 capsule a day).
  Synbiotic: The synbiotic to be used is fructo-oligosaccharide with a degree of polymerization < 10 at 4 g/twice a day (two sticks a day) plus Bifidobacterium animalis subsp. lactis BB-12 as minimum of 10 billion CFU/day (1 capsule a day).
- Total: Total of all reporting groups
Arm/Group | Synbiotic | Maltodextrin | Total
Number analyzed (Participants) | 45 | 44 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (12.4) | 51.6 (13.1) | 50.8 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 31
  Male | 31 | 27 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 45 | 44 | 89
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 45 | 44 | 89
percentage liver fat [Median (Inter-Quartile Range); unit: percentage] — This data reflects data collected at the Baseline time point. Liver fat percentage is calculated from magnetic resonance spectroscopy imaging. The percentage of liver fat is calculated from the peak measurement of lipid. Values are recorded on a scale from 0% (no liver fat) to 100% (high liver fat).
  percentage | 26.9 [9.7 to 38.4] | 22.9 [12.9 to 44.7] | 25 [24.6 to 36.7]
ELF score [Mean (Standard Deviation); unit: units on a scale] — This data reflects data collected at the Baseline time point. The ELF Score is a liver fibrosis score that is calculated by use of an algorithm: ELF score score = -7.412 + (ln(HA)*0.681) + (ln(P3NP)*0.775) + (ln(TIMP1)*0.494).
  HA=hyaluronic acid concentration P3NP=procollagen 3 amino terminal peptide concentration TIMP1=tissue inhibitor matrix metalloproteinase 1 concentration. All are measured in serum.
  Low scores <7.7 are good for excluding fibrosis. High scores >9.8 are good for identifying fibrosis.
  units on a scale | 6.9 (0.4) | 6.9 (0.3) | 6.9 (0.4)
NAFLD fibrosis score [Mean (Standard Deviation); unit: units on a scale] — This data reflects data collected at the Baseline time point. NAFLD fibrosis score (NFS) is calculated using the following algorithm: -1.675 +0.037 ×age (years) +0.094 ×BMI (kg/m2) +1.13 × impaired fasting glucose (IFG)/diabetes (yes=1, no=0) +0.99 × aspartate aminotransferase (AST)/ alanine aminotransferase (ALT) ratio -0.013 ×platelet (×109/l) -0.66 ×albumin (g/dl).
  The score is used to classify the probability of fibrosis. A scores < -1.5 indicates a low probability, > -1.5 to < 0.67 indicates intermediate probability, and a score of > 0.67 indicates a high probability of liver fibrosis.
  units on a scale | -1.3 (1.3) | -1.2 (1.3) | -1.2 (1.3)
Bifidobacterium spp. [Median (Inter-Quartile Range); unit: percentage] — This data reflects data collected at the Baseline time point. Total bacteria and Bifidobacterium spp. were quantified using quantitative polymerase chain reaction (qPCR). The percentage of Bifidobacteria spp was computed as the percent of Bifidobacteria spp and the denominator was the total number of all bacteria.
  percentage | 0.8 [0.3 to 2.0] | 0.6 [0.1 to 1.9] | 0.8 [0.2 to 2.0]

OUTCOME MEASURES:

1. Primary Outcome: Change in Liver Fat
Description: Change in liver fat percent was calculated as the percent liver fat at the end of the study, minus the percent of liver fat prior to the intervention. Change in liver fat percent ranged from -60.6% (good) to + 33.7% (bad).
Time Frame: baseline and 12 months
Population: numerical difference between baseline measurement and 12 month measurement
Measure: Mean (95% Confidence Interval); unit: percentage of liver fat
Arm/Group | Synbiotic | Maltodextrin
Number analyzed (Participants) | 45 | 44
percentage of liver fat | -3.8 [-7.98 to 0.38] | -6.0 [-10.6 to -1.45]
Statistical Analysis 1: Comparison: Synbiotic vs Maltodextrin; A total sample size of 100 participants, with a 14% drop out during the study and 43 participants in each group completing the study provided 85% power to detect a difference of 40% in liver fat (in the treatment arm compared with the placebo), using a power calculation test with a 0.05 two-sided significance level. For change in liver fat percentage (and other secondary outcomes), ANCOVA will also be undertaken to assess effect sizes in the intervention group and placebo; Test type: Superiority; p = 0.05, Regression, Linear — The threshold for statistical significance was p=0.05; Mean Difference (Net) = -3.8, Standard Deviation 0.8
Statistical Analysis 2: Comparison: Synbiotic vs Maltodextrin; Test type: Superiority — For each primary outcome, a change variable was calculated as the difference between end of study and baseline measurements. Multiple regression analysis was used to assess the effect of synbiotic treatment on each of the change variables of interest; p < 0.001, Regression, Linear; Median Difference (Final Values) = -1.7

2. Primary Outcome: Change in Enhanced Liver Fibrosis Score (ELF)
Description: Change in Enhanced Liver Fibrosis score (ELF) was calculated as ELF score at the end of the study minus ELF score prior to the intervention (at baseline). A decrease in the ELF score was considered good as it reflected a decrease in liver fibrosis, and an increase in ELF score was considered bad as it reflected an increase in liver fibrosis.
  Change in ELF scores ranged from -0.56 (good) to + 0.68 (bad).
Time Frame: baseline and 12 months
Population: numerical difference between baseline measurement and 12 month measurement
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Synbiotic | Maltodextrin
Number analyzed (Participants) | 45 | 44
units on a scale | 0.12 [0.03 to 0.19] | 0.13 [0.05 to 0.19]
Statistical Analysis 1: Comparison: Synbiotic vs Maltodextrin; Test type: Superiority — For each primary outcome, a change variable was calculated as the difference between end-of study and baseline measurements. Multiple regression analysis was used to assess the effect of synbiotic treatment on each of the change variables of interest; p = 1.00, Regression, Linear; Mean Difference (Final Values) = 0.1

3. Primary Outcome: Change in NAFLD Fibrosis Score
Description: Change in NAFLD Fibrosis Score (NFS) was calculated as the NFS score at the end of the study, minus NFS score prior to the intervention (at baseline). A decrease in the NFS score was considered good because it reflected a decrease in liver fibrosis, and an increase in NFS score was considered bad, as it reflected an increase in liver fibrosis.
  Change in NFS scores ranged from -2.07 (good) to + 1.75 (bad)
Time Frame: baseline and 12 months
Population: numerical difference between baseline measurement and 12 month measurement
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Synbiotic | Maltodextrin
Number analyzed (Participants) | 45 | 44
units on a scale | -1.3 [-1.68 to -0.92] | -1.2 [-1.58 to -0.82]
Statistical Analysis 1: Comparison: Synbiotic vs Maltodextrin; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.80, Regression, Linear; Mean Difference (Final Values) = 0.2

4. Primary Outcome: Change in Bifidobacterium Spp.
Description: The change in percent of Bifidobacteria spp was computed as the percent of Bifidobactera spp at the end of the study minus the percent of Bifidobacteria prior to the intervention (at baseline).
  A positive change in percent (e.g +0.1 to 7.0%) in Bifidobacteria spp. was considered good and a negative change in percent (e.g. -0.1 to -0.5%) in Bifidobacteria spp. considered bad. (Minimum = -0.5% (bad) and Maximum = +7.0% (good)).
Time Frame: baseline and 12 months
Population: numerical difference between baseline measurement and 12 month measurement
Measure: Mean (95% Confidence Interval); unit: percentage of fecal Bifidobacterium spp
Arm/Group | Synbiotic | Maltodextrin
Number analyzed (Participants) | 45 | 44
percentage of fecal Bifidobacterium spp | 1.72 [0.89 to 2.55] | -0.02 [-0.46 to 0.42]
Statistical Analysis 1: Comparison: Synbiotic vs Maltodextrin; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Beta-diversity indexes; Beta-diversity indexes were first visualized through a Principal Coordinates Analysis (PCoA); Median Difference (Final Values) = 0.97

ADVERSE EVENTS:
Time Frame: The adverse event data were collected over the period of the study between baseline and end of study (total period 12 months).
Description: We used the clinicaltrials.gov definition for adverse event and/or serious adverse event.
Arm/Group | Synbiotic | Maltodextrin
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/49
Serious Adverse Events (participants affected / at risk) | 6/55 | 6/49
Other Adverse Events (participants affected / at risk) | 35/55 | 30/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Synbiotic (N=55) | Maltodextrin (N=49)
Back pain after Liver biopsy (Investigations) | 0 | 1
myocardial infarction (Cardiac disorders) | 0 | 1
abdominal pain, surgery (General disorders) | 2 | 2
breast cancer (Reproductive system and breast disorders) | 1 | 0
orthopedic (Musculoskeletal and connective tissue disorders) | 3 | 2
urinary tract cancer (Renal and urinary disorders) | 1 | 0
Hypertension (General disorders) | 0 | 1
chest infection (Respiratory, thoracic and mediastinal disorders) | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Synbiotic (N=55) | Maltodextrin (N=49)
Post adipose tissue biopsy pain (Surgical and medical procedures) | 2 | 2
diverticulosis, intestinal disorders (Gastrointestinal disorders) | 3 | 3
Nausea, vomitting and diarrhea (Gastrointestinal disorders) | 12 | 10
Headache, collapse, dizziness (General disorders) | 5 | 6
Flu, chest infection (Respiratory, thoracic and mediastinal disorders) | 14 | 13
dermatological problems (Skin and subcutaneous tissue disorders) | 2 | 1
dental problems (General disorders) | 4 | 1
anxiety and depression (General disorders) | 1 | 4
Liver alteration other than NAFLD (Hepatobiliary disorders) | 2 | 1
Joint pain, back pain (Musculoskeletal and connective tissue disorders) | 19 | 16
Skin infection, abrasion, rash (Skin and subcutaneous tissue disorders) | 8 | 7
urinary tract disorders (Renal and urinary disorders) | 7 | 1
chest pain, alterations on ecg (Cardiac disorders) | 3 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
vascular disorders (Vascular disorders) | 1 | 1
otorhinolaryngological disorders (Ear and labyrinth disorders) | 2 | 1
hypertension (General disorders) | 0 | 1
breast disorders (Reproductive system and breast disorders) | 1 | 0
nutrient deficiency (Metabolism and nutrition disorders) | 1 | 0
ophtalmology disorders (Eye disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
We choose one strain of bacteria in the synbiotic. The study was designed as a phase-2 clinical trial using magnetic resonance spectroscopy (MRS) and not liver biopsy. We deliberately did not include a lifestyle intervention as we wanted to test the effect of the synbiotic alone.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2014-07-31): https://cdn.clinicaltrials.gov/large-docs/40/NCT01680640/Prot_000.pdf
  • Statistical Analysis Plan (2014-06-04): https://cdn.clinicaltrials.gov/large-docs/40/NCT01680640/SAP_001.pdf